CLINICAL TRIAL: NCT05145426
Title: Investigation of Low-intensity Focused Ultrasound for Human Pain Management
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Wynn Legon, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21-796
Record Dates: First submitted 2021-11-10; First posted 2021-12-06 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-02

CONDITIONS: Chronic Pain
Keywords: Low-intensity focused ultrasound
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Multiple subject repeated measures
Masking Description: Sham trials will be utilized within subject. All subjects will receive sham and ultrasound conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain Trials (Experimental): Multi visit - LIFU/Sham application, with quantitative sensory testing (using peltier device).
  Interventions: Device: Low Intensity Focused Ultrasound

INTERVENTIONS:
Device: Low Intensity Focused Ultrasound — Application of LIFU

SUMMARY:
This project examines the effects of noninvasive brain stimulation on pain. The investigators believe this study will help to better understand possible treatments for chronic pain patients. Participants undergo structural imaging, a functional Magnetic Resonance Image (fMRI) and computed tomography (CT). These images are used to align the low-intensity focused ultrasound (LIFU) device which uses sound waves to temporarily change brain activity. Pain testing is done using a small device that will increase/decrease the temperature of the skin. Brain signals are collected using electroencephalography (EEG). Heart rate, blood pressure, and skin moisture will be monitored as well.

ELIGIBILITY:
Inclusion Criteria:

* Understand and speak English

Exclusion Criteria:

* MRI/CT/EEG contraindications.

  1. Claustrophobia
  2. Contraindications to MRI: including pacemaker, aneurysm clips, neurostimulators, cochlear implants, metal in eyes, steel worker, or other implants.
  3. Contraindications to CT: pregnancy
  4. Active medical disorder or treatment with potential CNS effects
  5. History of neurologic disorder
  6. History of head injury resulting in loss of consciousness for >10 minutes.
  7. History of alcohol or drug dependence
  8. Failure to provide Social Security Number or Tax ID number. This is required for tax purposes or payment cannot be processed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Perceived sensation score | Assessed per participant, over the course of participation - an average of 3 weeks.
  Changed perceived sensation score on a 1-10 scale in response to painful stimuli.

SECONDARY OUTCOMES:
Windup Pain | Assessed per participant, over the course of participation - an average of 3 weeks
  Changed windup pain score on a 1-10 scale.
CHEP Amplitude | Assessed per participant, over the course of participation - an average of 3 weeks
  Attenuated N1/P1 CHEP amplitude recorded with EEG

CONTACTS AND LOCATIONS:
Locations (1):
- Fralin Biomedical Research Institute, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Legon W, Sato TF, Opitz A, Mueller J, Barbour A, Williams A, Tyler WJ. Transcranial focused ultrasound modulates the activity of primary somatosensory cortex in humans. Nat Neurosci. 2014 Feb;17(2):322-9. doi: 10.1038/nn.3620. Epub 2014 Jan 12. PMID 24413698
- [Background] Tyler WJ. Noninvasive neuromodulation with ultrasound? A continuum mechanics hypothesis. Neuroscientist. 2011 Feb;17(1):25-36. doi: 10.1177/1073858409348066. Epub 2010 Jan 25. PMID 20103504
- [Background] Kubanek J, Shukla P, Das A, Baccus SA, Goodman MB. Ultrasound Elicits Behavioral Responses through Mechanical Effects on Neurons and Ion Channels in a Simple Nervous System. J Neurosci. 2018 Mar 21;38(12):3081-3091. doi: 10.1523/JNEUROSCI.1458-17.2018. Epub 2018 Feb 20. PMID 29463641
- [Background] Kamimura HA, Wang S, Chen H, Wang Q, Aurup C, Acosta C, Carneiro AA, Konofagou EE. Focused ultrasound neuromodulation of cortical and subcortical brain structures using 1.9 MHz. Med Phys. 2016 Oct;43(10):5730. doi: 10.1118/1.4963208. PMID 27782686
- [Derived] Legon W, Strohman A, In A, Payne B. Noninvasive neuromodulation of subregions of the human insula differentially affect pain processing and heart-rate variability: a within-subjects pseudo-randomized trial. Pain. 2024 Jul 1;165(7):1625-1641. doi: 10.1097/j.pain.0000000000003171. Epub 2024 Feb 1. PMID 38314779